CLINICAL TRIAL: NCT04237012
Title: Randomized Self-Controlled Treatment With an Intracanalicular Dexamethasone Insert Compared to Topical Over the Counter Lubrication Therapy in Patients With Bilateral Ocular Surface Disease
Brief Title: ACCURATE Study for Subjects With Dry Eyes
Acronym: ACCURATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Eye Centers of Racine and Kenosha (Other)
Responsible Party: Principal Investigator, Inder Paul Singh, M.D., I. Paul Singh, M.D. Principal Investigator, The Eye Centers of Racine and Kenosha
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WIRB Protocol # 20192595
Record Dates: First submitted 2020-01-13; First posted 2020-01-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dextenza (Experimental): Treatment Arm-Dextenza insertion lower lid punctum at time of screening and use of OTC artificial tears as needed
  Interventions: Drug: Dextenza 0.4Mg Intracanalicular Insert
- Over the counter Artificial tears (Active Comparator): Controlled arm: continuation of OTC artificial tears no placement of Dextenza intracanular insert
  Interventions: Other: Over the counter Artificial tears

INTERVENTIONS:
Drug: Dextenza 0.4Mg Intracanalicular Insert — all patients will receive Intracanalicular dexamethasone, 0.4mg insert lower punctum and able to use over the counter artificial tears PRN at patient discretion
  Other Names: dexamethasone
  Arms: Dextenza
Other: Over the counter Artificial tears — over the counter artificial tears PRN at patient discretion
  Arms: Over the counter Artificial tears

SUMMARY:
To determine treatment and imaging outcomes in bilateral ocular surface disease management with an intracanalicular dexamethasone (0.4 mg) insert compared to standard topical over-the-counter artificial tears lubrication management

DETAILED DESCRIPTION:
This study will evaluate the benefit of treatment with a physician administered intracanalicular dexamethasone insert and patient administered artificial tears prn compared to patient administered artificial tears prn (control) in patients with bilateral ocular surface dry eye disease. The study is a self-controlled design and includes multiple objective, measureable, and quantifiable endpoints to best determine an objective response to treatment in patient eyes randomized to either the insert plus prn artificial tears or artificial tears prn control. To aid in ensuring best possible masking, DEXTENZA is best visualized with blue light and yellow filter and therefore visualization will not be assessed until final visit following all measures.

ELIGIBILITY:
Inclusion Criteria:A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* Age 18 years and older
* Demonstrate objective signs of Ocular Surface Disease (OSD) or
* Demonstrate symptoms of OSD determined by a standardized questionnaire
* No other corneal pathology to create unknown variability

Exclusion Criteria:A patient who meets any of the following criteria in either eye will be excluded from the study:

* History of using topical steroids or other anti-inflammatory drops within 6 months of the study
* History of corticosteroid implant (Ozurdex or Iluvien) or intravitreal steroid use for macular disease in last 12 months
* History or current use of oral steroids or immunosuppressants
* Active ocular infection
* History of HSV
* History corneal refractive surgery
* Uncontrolled Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Determine effect of dexamethasone insert over artificial tears | 1 month
  To determine the effect of dexamethasone insert plus over-the-counter artificial tears prn compared to over the counter artificial tears prn from Baseline at Week 2 (at 8 am, 12 pm and 4 pm) as measured by iTrace and IOL Master 700: and comfort of dry eyes using the OSDI scale and reading scores

SECONDARY OUTCOMES:
OSDI scores | 1 month
  comfort of dry eyes using the OSDI scale and reading scores, scores are from the SPEED questionnaire. scale from 0-3 0-Never 1- Sometime 2-Often 3-Constant for the symptoms

OTHER OUTCOMES:
ITRACE | 1 month
  measured by iTrace to measure comfort of dry eyes, no scale just review the changes if there are any
IOL Master | 1 month
  as measured by IOL Master 700 to measure comfort of dry eyes, compare the previous images after each visit

CONTACTS AND LOCATIONS:
Overall Officials: Inder P Singh, M.D., Principal Investigator — President
Locations (1):
- The Eye Center of Racine, Racine, Wisconsin, United States